CLINICAL TRIAL: NCT04056234
Title: Study of the Articular Microbiota in Rheumatoid Arthritis.
Acronym: MICROPORE
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHU BX 2011/12
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Rheumatoid Arthritis; Synovial Disorder; Arthrosis
Keywords: Translocation; Synovial microbiota
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis | interventions — Arthrocentesis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The joint fluid samples will be obtained from residues of samples taken for diagnostic or therapeutic purposes.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rheumatoid arthritis group: Patients with rheumatoid arthritis
  Interventions: Procedure: Joint puncture
- Control group: Patients with osteoarthritis / joint effusion.
  Interventions: Procedure: Joint puncture

INTERVENTIONS:
Procedure: Joint puncture — Patient requiring joint puncture for diagnostic or therapeutic reasons.

SUMMARY:
The cause of rheumatoid arthritis (RA) remains unknown, although major advances have been done these last ten years in the comprehension of its pathophysiology.

The aim of this study is to described a synovial microbiota specific for rheumatoid arthritis.

DETAILED DESCRIPTION:
The cause of rheumatoid arthritis (RA) remains unknown, although major advances have been done these last ten years in the comprehension of its pathophysiology. One of the most significant discoveries was the post-translational modification of various self-proteins resulting in the replacement of arginine residues by citrulline. This conversion results in modifications of the basic charge of the peptides, of its primary and secondary structure, and the transformed peptides can then bound to some HLA-DR molecules (HLA-DR4, HLA-DR1), that are the best well known genetic factors of rheumatoid arthritis (RA). This leads to immunization to citrullinated peptides in genetically predisposed patients, which is now identified as the most characteristic auto-immun phenomenon of RA. Anti-citrullinated peptide antibodies (ACPA) have become the most relevant biologic test for the diagnosis of RA.

The conversion to citrulline is due to the action of an enzyme, the peptidyl arginine deiminase (PAD). Endogenous PADs have been identified in humans, but their activation needs high concentrations of calcium in the cells that are not physiological. Thus, the activation of self-PADs occurs only in extreme conditions, such as apoptosis, or major stresses resulting from toxic or infectious process. But some bacteria also contain PADs that are involved in their energetic metabolism. Two main factors have yet been identified to lead to citrullination of self-peptides and are now recognized as important environment risk factors for RA: smoking and periodontitis. Periodontitis is the consequence of an infection that is mainly due to Porphyromonas gingivalis, one of the bacteria processing a PAD. These facts reinforce the old hypothesis of an infectious origin of RA.

However, all RA patients are neither smoker nor affected by periodontitis, and many other bacteria have PADs and may be involved in the pathophysiology of RA. Moreover, it has been demonstrated that citrullination process and ACPA production can precede RA for years, while the citrullination and ACPA production are located to a mucous membrane (oral, pulmonary…). How these processes reach the joint remains a mystery.

The hypothesis is that the involved bacteria translocate to the joint, inducing local citrullination of synovial peptides, inflammation and production of ACPA within the joint, and resulting in arthritis.

The aim of this study is to demonstrate this translocation of bacteria in the synovium, and to described a synovial microbiota specific for rheumatoid arthritis .

Pilot study, including only few patients, just to demonstrate the validity of the translocation concept and the performance of the procedures.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting with RA according to ACR87 and ACR/EULAR 2010 criteria
* patients presenting with RA anti-citrullinated peptide antibodies positive
* patients presenting with active RA, characterized by at least one synovitis
* patients presenting with an arthritis requiring arthrocentesis and synovial fluid collection for diagnostic or therapeutic purpose
* patients giving agreement to participate to the study and to sign informed consent.

Exclusion Criteria:

* patients suffering from osteoarthritis
* patients presenting with joint effusion justifying an arthrocentesis and synovial fluid collection for diagnostic of therapeutic purpose
* patients giving agreement to participate to the study and to sign informed consent
* Patients presenting with another arthropathy than anti-citrullinated peptide antibodies positive RA or osteoarthritis
* Patients not requiring arthrocentesis for medical reasons
* Patients refusing to sign informed consent
* Patients presenting with understanding problems due to language or cognitive reasons.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a pilot study. The number of subjets will be 12 RA patients and 6 controls suffering from osteoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2012-02-21 (Actual); Primary Completion 2013-02-22 (Actual); Study Completion 2013-02-22 (Actual)

PRIMARY OUTCOMES:
Presence of bacterial DNA by 16s PCR | At the screening
  Detection by 16s PCR of DNA of bacterial origin in synovial fluid specimens
Presence of a characteristic microbiota | At the screening
  Research of a characteristic microbiota of rheumatoid arthritis

CONTACTS AND LOCATIONS:
Overall Officials: Emilie SHIPLEY, Dr, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No